CLINICAL TRIAL: NCT03958214
Title: Promoting Self-Regulation Skills and Healthy Eating Habits in Early Head Start
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Penn State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2016-0465; A271000 (Other: UW Madison); SOHE/SOHE/SOHE*ADMIN (Other: UW Madison)
Record Dates: First submitted 2017-02-11; First posted 2019-05-21 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Poverty

STUDY DESIGN:
Intervention Model Description: Families are blocked within home visitor caseload and randomly assigned to receive the new curriculum or usual practice Early Head Start home visits for 12 weeks.
Who Masked: Outcomes Assessor
Masking Description: All interviews are conducted by research assistants who are blind to study condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recipe 4 Success (Experimental): For 12 weeks, home visitors will stop delivering the usual practice Early Head Start home visits and deliver the Recipe 4 Success curriculum instead. At the end of 12 weeks, home visitors will resume usual practice Early Head Start home visits.
  Interventions: Behavioral: Recipe 4 Success
- Usual practice Early Head Start (Active Comparator): Home visitors will continue to deliver usual practice Early Head Start home visits that follow a standard curriculum and are tailored on an ongoing basis to meet individual family needs.
  Interventions: Behavioral: Usual practice Early Head Start

INTERVENTIONS:
Behavioral: Recipe 4 Success — Home visitors teach parents about children's self-regulation skills and healthy eating habits. The home visitors then teach parents how to sensitively scaffold the development of their toddlers' self-regulation skills in the context of cooking and snack preparation lessons. Prior research shows that self-regulation skills in early childhood predict long-term health indicators, such as BMI. Prior research also shows that children who are involved in the preparation of healthier foods are more likely to eat them.
  Arms: Recipe 4 Success
Behavioral: Usual practice Early Head Start — Home visitors will continue to deliver usual practice Early Head Start home visits that follow a standard curriculum and are tailored on an ongoing basis to meet individual family needs.
  Arms: Usual practice Early Head Start

SUMMARY:
The purpose of this study is to test the effectiveness of a new curriculum on toddlers' self-regulation skills and healthy eating habits. The curriculum is being delivered as part of Early Head Start home visits and compared to the effectiveness of usual practice Early Head Start home visits.

ELIGIBILITY:
Inclusion Criteria:

* Children must be receiving Early Head Start home visits and be at least 2 years old at the beginning of the study.

Exclusion Criteria:

-

Ages: 2 Years to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 244 (Actual)
Dates: Start 2016-11-08 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Change in children's healthy eating habits: Body mass index | Baseline / up to 18 months
  Healthy eating habits will be assessed through change in body mass index
Change in children's healthy eating habits: Food diaries | Baseline / up to 18 months
  Healthy eating habits will be assessed through change in consumption of fruits/vegetables and junk food, as assessed with 24-hour food diaries
Change in children's healthy eating habits: Parent reports | Baseline / up to 18 months
  Healthy eating habits will be assessed through parent survey of pickiness, etc.; mean scores reported from 5-point Likert scales with higher scores indicating healthier eating habits
Change in children's self-control skills: Direct testing | Baseline / up to 18 months
  Children's self-control skills will be assessed through direct testing (e.g., snack delay task)
Change in children's self-control skills: Video interactions | Baseline / up to 18 months
  Children's self-control skills will be assessed through parent-child interactions, rated on Likert scale from video recordings; mean score reported between 1 = almost never and 5 = almost always
Change in children's self-control skills: Parent ratings | Baseline / up to 18 months
  Children's self-control skills will be assessed through parent ratings on standardized behavior checklists; mean scores reported from 3- or 5-point Likert scales with higher scores indicating greater self-control
Change in parents' sensitive/responsiveness: Video interactions | Baseline / up to 18 months
  Parents' sensitive/responsiveness will be assessed through parent-child interactions, rated on Likert scale from video recordings; mean score reported between 1 = almost never and 5 = almost always
Change in parents' sensitive/responsiveness: Parent ratings | Baseline / up to 18 months
  Parents' sensitive/responsiveness will be assessed through parent ratings on standardized surveys; mean scores reported from 5-point Likert scales with higher scores indicating greater sensitive/responsiveness

SECONDARY OUTCOMES:
Change in children's sleep habits: Parent reports | Baseline / up to 18 months
  Sleep habits will be assessed through parent survey; mean scores reported from 5-point Likert scales with higher scores indicating better sleep habits

CONTACTS AND LOCATIONS:
Overall Officials: Robert Nix, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Engbretson AM, Nix RL, Park YR, Gill S, Hostetler ML. Elaboration of parents' schemas of their children: Unique relations to sensitivity and learning support among families living in poverty. J Fam Psychol. 2023 Apr;37(3):318-323. doi: 10.1037/fam0001048. Epub 2023 Jan 2. PMID 36595449